CLINICAL TRIAL: NCT01723254
Title: A Phase 1, Randomized, Double Blinded, Placebo Controlled Study To Evaluate The Safety, Tolerability, Immunogenicity, And Exploratory Pharmacodynamic Response Of Ascending Dose Levels Of An Anti-ige Vaccine With Two Different Adjuvant Formulations (Pf-06444753 And Pf-06444752) In Generally Healthy Subjects With Allergic Rhinitis
Brief Title: A Study To Assess The Safety And Tolerability Of Different Doses Of PF-06444753 And PF-06444752 In Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B4901001; ANTI- IGE VACCINE (Other: Alias Study Number)
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Allergic Rhinitis
Keywords: Vaccines; Phase 1; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-06444753 (Experimental)
  Interventions: Biological: IGE-1
- PF-06444752 (Experimental)
  Interventions: Biological: IGE-2
- Placebo (Placebo Comparator): Intramuscular
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: IGE-1 — Intramuscular, multiple dose
  Arms: PF-06444753
Biological: IGE-2 — Intramuscular, multiple dose
  Arms: PF-06444752
Biological: Saline — Saline (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of different doses of PF-06444753 and PF-06444752 in subjects with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, males or females of non-child bearing potential, who are between 18 and 55 years, inclusive,
* Intermittent or persistent allergic rhinitis that is associated with perennial or seasonal allergen reactivity at screening as determined by a positive specific IgE level ≥1 KU/L to at least one of the following common allergens: dust mite (Dermatophagoides farinae or Dermatophagoides pteronyssinus), cat, dog, mold (Alternaria), Bermuda grass, common ragweed, oak, Timothy grass or elm.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease that may compromise their ability to safely participate in the study.
* Evidence or history of clinically significant pulmonary disease (including allergic and non-allergic asthma, chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis, chronic bronchitis, emphysema, tuberculosis, pulmonary fibrosis, pulmonary hypertension, or others).
* Evidence or history of clinically significant autoimmune disease (including rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, or others).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Canada (4):
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Diex Research Montreal Inc., Montreal, Quebec
  - Centre de Recherche Appliquee en Allergie de Quebec, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4901001&StudyName=A%20Study%20To%20Assess%20The%20Safety%20And%20Tolerability%20Of%20Different%20Doses%20Of%20PF-06444753%20And%20PF-06444752%20In%20Subjects%20With%20Allergic%20Rhinitis

RESULTS

PARTICIPANT FLOW:
Groups:
- IGE-1 6 mcg: Participants received study vaccine IGE-1 (PF-06444753) 6 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-1 20 mcg: Participants received study vaccine IGE-1 (PF-06444753) 20 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-1 60 mcg: Participants received study vaccine IGE-1 (PF-06444753) 60 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-1 200 mcg: Participants received study vaccine IGE-1 (PF-06444753) 200 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-2 20 mcg: Participants received study vaccine IGE-2 (PF-06444752) 20 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-2 60 mcg: Participants received study vaccine IGE-2 (PF-06444752) 60 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- IGE-2 200 mcg: Participants received study vaccine IGE-2 (PF-06444752) 200 micrograms (mcg) on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a toll-like receptor 9 [TLR9] agonist) in combination as adjuvants.
- Saline Placebo: Participants received saline placebo matching IGE-1 or IGE-2 on Days 1, 28, 56, and 168. Placebo was also administered intramuscularly in the upper deltoid muscle on the participant's preferred side.
Period: Overall Study
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Started | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63
Completed | 5 | 18 | 17 | 18 | 18 | 18 | 19 | 60
Not Completed | 1 | 3 | 3 | 2 | 2 | 2 | 1 | 3
Not completed — Conflict with work schedule | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Personal issues | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No longer have time to participate | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Move/Left to another country/city | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo | Total
Number analyzed (Participants) | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (13.3) | 31.6 (8.8) | 35.7 (10.0) | 33.5 (9.3) | 35.4 (9.2) | 35.9 (11.0) | 33.6 (12.0) | 34.7 (8.8) | 34.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 5 | 10
  Male | 6 | 21 | 19 | 19 | 19 | 18 | 20 | 58 | 180

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants With Local Reactions By Severity Within 14 Days of Any Vaccination
Description: Local reactions consisted of any pain at the site of injection, any swelling, and any redness. Participants were issued an electronic diary (e-diary) and were asked to monitor and record (according to corresponding grading scales) any local reactions for 14 days following each vaccination. Grading details are as follows: Mild (Pain: did not interfere with activity; Redness and Swelling: 0.5-5.0 centimeters [cm] or 1-10 caliper units), Moderate (Pain: interfered with activity; Redness and Swelling: more than [>] 5.0 to 10.0 cm or 11-20 caliper units), Severe (Pain: prevented daily activity; Redness and Swelling: >10 cm or 21 caliper units and above).
Time Frame: Within 14 days
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Groups:
- IGE-1 6 mcg: Participants received study vaccine IGE-1 (PF-06444753) 6 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-1 20 mcg: Participants received study vaccine IGE-1 (PF-06444753) 20 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-1 60 mcg: Participants received study vaccine IGE-1 (PF-06444753) 60 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-1 200 mcg: Participants received study vaccine IGE-1 (PF-06444753) 200 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-1 and IGE-2 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-2 20 mcg: Participants received study vaccine IGE-2 (PF-06444752) 20 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-2 60 mcg: Participants received study vaccine IGE-2 (PF-06444752) 60 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
- IGE-2 200 mcg: Participants received study vaccine IGE-2 (PF-06444752) 200 mcg on Days 1, 28, 56, and 168. Study vaccine volume was 0.5 mL and was administered intramuscularly in the upper deltoid muscle on the participant's preferred side. IGE-2 and IGE-1 contained the same antigenic material but differed in their fixed adjuvant configurations: IGE-1 was with aluminum hydroxide (alum) alone and IGE-2 with alum and CpG 24555 (CpG; a TLR9 agonist) in combination as adjuvants.
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Number analyzed (Participants) | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63
Percentage of participants
  Any Redness | 50.0 [20.1 to 79.9] | 9.5 [2.6 to 23.4] | 30.0 [16.6 to 46.7] | 15.0 [5.6 to 30.4] | 20.0 [9.0 to 36.1] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 7.9 [3.9 to 14.2]
  Mild Redness | 50.0 [20.1 to 79.9] | 9.5 [2.6 to 23.4] | 30.0 [16.6 to 46.7] | 15.0 [5.6 to 30.4] | 20.0 [9.0 to 36.1] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 7.9 [3.9 to 14.2]
  Moderate and Severe Redness | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Any Swelling | 16.7 [1.7 to 51.0] | 14.3 [5.4 to 29.1] | 20.0 [9.0 to 36.1] | 30.0 [16.6 to 46.7] | 15.0 [5.6 to 30.4] | 5.0 [0.5 to 18.1] | 5.0 [0.5 to 18.1] | 9.5 [5.1 to 16.1]
  Mild Swelling | 16.7 [1.7 to 51.0] | 14.3 [5.4 to 29.1] | 15.0 [5.6 to 30.4] | 20.0 [9.0 to 36.1] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 5.0 [0.5 to 18.1] | 9.5 [5.1 to 16.1]
  Moderate Swelling | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Severe Swelling | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Pain | 83.3 [49.0 to 98.3] | 100.0 [89.6 to 100.0] | 90.0 [75.5 to 97.3] | 100.0 [89.1 to 100.0] | 90.0 [75.5 to 97.3] | 85.0 [69.6 to 94.4] | 90.0 [75.5 to 97.3] | 15.9 [10.1 to 23.4]
  Mild Pain | 50.0 [20.1 to 79.9] | 57.1 [41.0 to 72.2] | 50.0 [33.8 to 66.2] | 20.0 [9.0 to 36.1] | 80.0 [63.9 to 91.0] | 75.0 [58.5 to 87.3] | 60.0 [43.3 to 75.1] | 14.3 [8.8 to 21.6]
  Moderate Pain | 33.3 [9.3 to 66.7] | 38.1 [23.6 to 54.4] | 40.0 [24.9 to 56.7] | 70.0 [53.3 to 83.4] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 30.0 [16.6 to 46.7] | 1.6 [0.2 to 6.0]
  Severe Pain | 0.0 [0.0 to 31.9] | 4.8 [0.5 to 17.3] | 0.0 [0.0 to 10.9] | 10.0 [2.7 to 24.5] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Local Reaction | 83.3 [49.0 to 98.3] | 100.0 [89.6 to 100.0] | 90.0 [75.5 to 97.3] | 100.0 [89.1 to 100.0] | 95.0 [81.9 to 99.5] | 85.0 [69.6 to 94.4] | 90.0 [75.5 to 97.3] | 25.4 [18.3 to 33.8]
  Any Severe Local Reaction | 0.0 [0.0 to 31.9] | 4.8 [0.5 to 17.3] | 0.0 [0.0 to 10.9] | 10.0 [2.7 to 24.5] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]

2. Primary Outcome: Percentages of Participants With Systemic Reactions By Severity Within 14 Days of Any Vaccination
Description: Systemic reactions consisted of fever, vomiting, diarrhea, headache, fatigue, muscle pain (other than at the injection site) and joint pain (other than pain adjacent to injection site). Participants were issued an electronic diary (e-diary) and were asked to monitor and record (according to corresponding grading scales) any systemic reactions for 14 days following each vaccination. Grading details are as follows: Mild (Vomiting: 1-2 times in 24 hours; Diarrhea: 2-3 loose stools in 24 hours; Headache, Fatigue, Muscle Pain, Joint Pain: no interference with activity), Moderate (Vomiting: >2 times in 24 hours; Diarrhea: 4-5 loose stools in 24 hours; Headache, Fatigue, Muscle and Joint Pain: some interference with activity), Severe (Vomiting: required intravenous hydration; Diarrhea: more than or equal to [>=] 6 stool in 24 hours; Headache, Fatigue, Muscle and Joint Pain: Significant, prevented daily activity).
Time Frame: Within 14 days
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Number analyzed (Participants) | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63
Percentage of participants
  Any Fever | 0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 10.0 [2.7 to 24.5] | 20.0 [9.0 to 36.1] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 25.0 [12.7 to 41.5] | 1.6 [0.2 to 6.0]
  Mild Fever | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 10.0 [2.7 to 24.5] | 15.0 [5.6 to 30.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 10.0 [2.7 to 24.5] | 1.6 [0.2 to 6.0]
  Moderate Fever | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 0.0 [0.0 to 3.6]
  Severe Fever | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 3.6]
  Any Vomiting | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 10.0 [2.7 to 24.5] | 10.0 [2.7 to 24.5] | 15.0 [5.6 to 30.4] | 0.0 [0.0 to 10.9] | 4.8 [1.8 to 10.3]
  Mild Vomiting | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 15.0 [5.6 to 30.4] | 0.0 [0.0 to 10.9] | 4.8 [1.8 to 10.3]
  Moderate Vomiting | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Severe Vomiting | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Diarrhea | 0.0 [0.0 to 31.9] | 47.6 [32.1 to 63.6] | 35.0 [20.7 to 51.8] | 55.0 [38.5 to 70.7] | 45.0 [29.3 to 61.5] | 30.0 [16.6 to 46.7] | 40.0 [24.9 to 56.7] | 42.9 [34.4 to 51.7]
  Mild Diarrhea | 0.0 [0.0 to 31.9] | 28.6 [15.8 to 44.8] | 25.0 [12.7 to 41.5] | 50.0 [33.8 to 66.2] | 30.0 [16.6 to 46.7] | 20.0 [9.0 to 36.1] | 30.0 [16.6 to 46.7] | 28.6 [21.1 to 37.1]
  Moderate Diarrhea | 0.0 [0.0 to 31.9] | 19.0 [8.6 to 34.5] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 10.0 [2.7 to 24.5] | 10.0 [2.7 to 24.5] | 14.3 [8.8 to 21.6]
  Severe Diarrhea | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Headache | 16.7 [1.7 to 51.0] | 81.0 [65.5 to 91.4] | 55.0 [38.5 to 70.7] | 70.0 [53.3 to 83.4] | 75.0 [58.5 to 87.3] | 60.0 [43.3 to 75.1] | 55.0 [38.5 to 70.7] | 65.1 [56.3 to 73.1]
  Mild Headache | 0.0 [0.0 to 31.9] | 47.6 [32.1 to 63.6] | 25.0 [12.7 to 41.5] | 40.0 [24.9 to 56.7] | 50.0 [33.8 to 66.2] | 30.0 [16.6 to 46.7] | 25.0 [12.7 to 41.5] | 39.7 [31.3 to 48.5]
  Moderate Headache | 16.7 [1.7 to 51.0] | 33.3 [19.6 to 49.7] | 30.0 [16.6 to 46.7] | 30.0 [16.6 to 46.7] | 25.0 [12.7 to 41.5] | 30.0 [16.6 to 46.7] | 30.0 [16.6 to 46.7] | 23.8 [16.9 to 32.1]
  Severe Headache | .0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 1.6 [0.2 to 6.0]
  Any Fatigue | 50.0 [20.1 to 79.9] | 61.9 [45.6 to 76.4] | 85.0 [69.6 to 94.4] | 85.0 [69.6 to 94.4] | 70.0 [53.3 to 83.4] | 60.0 [43.3 to 75.1] | 65.0 [48.2 to 79.3] | 66.7 [57.9 to 74.6]
  Mild Fatigue | 16.7 [1.7 to 51.0] | 19.0 [8.6 to 34.5] | 25.0 [12.7 to 41.5] | 35.0 [20.7 to 51.8] | 30.0 [16.6 to 46.7] | 35.0 [20.7 to 51.8] | 25.0 [12.7 to 41.5] | 23.8 [16.9 to 32.1]
  Moderate Fatigue | 33.3 [9.3 to 66.7] | 42.9 [27.8 to 59.0] | 55.0 [38.5 to 70.7] | 45.0 [29.3 to 61.5] | 40.0 [24.9 to 56.7] | 25.0 [12.7 to 41.5] | 40.0 [24.9 to 56.7] | 42.9 [34.4 to 51.7]
  Severe Fatigue | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 5.0 [0.5 to 18.1] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Muscle Pain | 66.7 [33.3 to 90.7] | 71.4 [55.2 to 84.2] | 75.0 [58.5 to 87.3] | 75.0 [58.5 to 87.3] | 70.0 [53.3 to 83.4] | 50.0 [33.8 to 66.2] | 60.0 [43.3 to 75.1] | 34.9 [26.9 to 43.7]
  Mild Muscle Pain | 33.3 [9.3 to 66.7] | 52.4 [36.4 to 67.9] | 45.0 [29.3 to 61.5] | 40.0 [24.9 to 56.7] | 45.0 [29.3 to 61.5] | 30.0 [16.6 to 46.7] | 25.0 [12.7 to 41.5] | 15.9 [10.1 to 23.4]
  Moderate Muscle Pain | 16.7 [1.7 to 51.0] | 19.0 [8.6 to 34.5] | 30.0 [16.6 to 46.7] | 35.0 [20.7 to 51.8] | 25.0 [12.7 to 41.5] | 20.0 [9.0 to 36.1] | 35.0 [20.7 to 51.8] | 19.0 [12.8 to 26.9]
  Severe Muscle Pain | 16.7 [1.7 to 51.0] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Joint Pain | 50.0 [20.1 to 79.9] | 33.3 [19.6 to 49.7] | 35.0 [20.7 to 51.8] | 35.0 [20.7 to 51.8] | 45.0 [29.3 to 61.5] | 35.0 [20.7 to 51.8] | 35.0 [20.7 to 51.8] | 20.6 [14.1 to 28.6]
  Mild Joint Pain | 33.3 [9.3 to 66.7] | 28.6 [15.8 to 44.8] | 20.0 [9.0 to 36.1] | 20.0 [9.0 to 36.1] | 35.0 [20.7 to 51.8] | 30.0 [16.6 to 46.7] | 25.0 [12.7 to 41.5] | 12.7 [7.5 to 19.8]
  Moderate Joint Pain | 16.7 [1.7 to 51.0] | 4.8 [0.5 to 17.3] | 15.0 [5.6 to 30.4] | 15.0 [5.6 to 30.4] | 10.0 [2.7 to 24.5] | 5.0 [0.5 to 18.1] | 10.0 [2.7 to 24.5] | 7.9 [3.9 to 14.2]
  Severe Joint Pain | 0.0 [0.0 to 31.9] | 0.0 [0.0 to 10.4] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 10.9] | 0.0 [0.0 to 3.6]
  Any Systemic Reaction | 66.7 [33.3 to 90.7] | 100.0 [89.6 to 100.0] | 90.0 [75.5 to 97.3] | 100.0 [89.1 to 100.0] | 95.0 [81.9 to 99.5] | 85.0 [69.6 to 94.4] | 85.0 [69.6 to 94.4] | 82.5 [74.8 to 88.6]
  Any Severe Systemic Reaction | 16.7 [1.7 to 51.0] | 0.0 [0.0 to 10.4] | 5.0 [0.5 to 18.1] | 5.0 [0.5 to 18.1] | 5.0 [0.5 to 18.1] | 0.0 [0.0 to 10.9] | 5.0 [0.5 to 18.1] | 1.6 [0.2 to 6.0]

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations From Treatment Due to TEAEs
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Severe TEAEs were those that interfered significantly with the participant's usual function. Causality assessment was made by the investigator.
Time Frame: Baseline up to 336 days post study administration or at Early Termination
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Number analyzed (Participants) | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63
participants
  Participants with TEAEs | 5 | 18 | 20 | 20 | 19 | 19 | 17 | 55
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Participants with severe TEAEs | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 4
  Permanent discontinuations due to TEAEs | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Temporary discontinuations due to TEAEs | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 4
  Participants with treatment-related TEAEs | 0 | 2 | 1 | 4 | 1 | 0 | 0 | 3

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, hormones, clinical chemistry, immunology urinalysis, urinalysis (dipstick and microscopy), and other tests such as human immunodeficiency virus antibody and hepatitis C antibody.
Time Frame: Baseline up to 336 days post last study drug administration or Early Termination
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Number analyzed (Participants) | 6 | 21 | 20 | 20 | 20 | 20 | 20 | 63
participants | 5 | 9 | 12 | 13 | 13 | 12 | 10 | 36

5. Secondary Outcome: Enzyme-Linked Immunosorbent Assay (ELISA) Measured Anti-IgE Geometric Mean Titers (GMTs) at Baseline, Day 182, and Day 336
Description: Ability of vaccine induced serum anti-immunoglobulin E (IgE) antibodies to interfere with IgE binding to recombinant alpha chain of the high affinity IgE receptor was assessed in an ELISA based assay. GMTs were calculated both as crude means (unadjusted) and by an analysis of covariance (ANCOVA) model with natural log transformed antibody titer as outcome variable, and treatment group as factor and baseline (in log scale) as covariates at each of the post dose measurement.
Time Frame: Baseline (Day 1), Day 182 (2 weeks after last vaccination), and end of study (Day 336)
Population: All randomized participants who received at least 1 dose of randomized treatment, n=number of evaluable participants at the specified time point.
Measure: Number (80% Confidence Interval); unit: units/milliliter (u/mL)
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Number analyzed (Participants) | 6 | 21 | 60 | 20 | 20 | 20 | 20 | 63
units/milliliter (u/mL)
  Day 1 (n=6,21,20,20,20,20,20,62) | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8] | 2002.8 [2002.8 to 2002.8]
  Day 182 (n=5,18,16,19,19,18,19,57) | 11310.6 [5642.0 to 22674.9] | 44480.1 [30845.9 to 64141.0] | 72925.4 [49484.3 to 107470.7] | 126981.7 [88942.3 to 181290.0] | 35833.4 [25031.3 to 51296.9] | 41947.5 [29086.0 to 60496.1] | 106036.8 [73954.8 to 152036.2] | 2147.9 [1745.8 to 2642.7]
  Day 336 (n=5,18,16,17,18,16,6,52) | 1896.7 [846.6 to 4248.9] | 17836.4 [11665.8 to 27271.1] | 22611.2 [14425.4 to 35442.0] | 42772.1 [27643.3 to 66180.7] | 9642.9 [6298.5 to 14763.1] | 12490.1 [7966.5 to 19582.1] | 43979.2 [20992.0 to 92138.2] | 2265.3 [1761.5 to 2913.2]

ADVERSE EVENTS:
Time Frame: Baseline up to 336 days post study administration or at Early Termination
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and a nonserious event during the study.
Arm/Group | IGE-1 6 mcg | IGE-1 20 mcg | IGE-1 60 mcg | IGE-1 200 mcg | IGE-2 20 mcg | IGE-2 60 mcg | IGE-2 200 mcg | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/21 | 0/20 | 0/20 | 0/20 | 1/20 | 0/20 | 1/63
Other Adverse Events (participants affected / at risk) | 5/6 | 17/21 | 20/20 | 20/20 | 19/20 | 19/20 | 17/20 | 54/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGE-1 6 mcg (N=6) | IGE-1 20 mcg (N=21) | IGE-1 60 mcg (N=20) | IGE-1 200 mcg (N=20) | IGE-2 20 mcg (N=20) | IGE-2 60 mcg (N=20) | IGE-2 200 mcg (N=20) | Saline Placebo (N=63)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IGE-1 6 mcg (N=6) | IGE-1 20 mcg (N=21) | IGE-1 60 mcg (N=20) | IGE-1 200 mcg (N=20) | IGE-2 20 mcg (N=20) | IGE-2 60 mcg (N=20) | IGE-2 200 mcg (N=20) | Saline Placebo (N=63)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 5 | 1 | 0 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 3
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 3
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 4 | 2 | 4 | 2 | 6 | 10
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 4
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 7 | 10 | 11 | 8 | 11 | 6 | 26
Vaginal infection (Infections and infestations) | 0/0 | 0/0 | 0/1 | 0/1 | 0/1 | 0/2 | 0/0 | 1/5 — Gender-specific event.
Vulvovaginitis (Infections and infestations) | 0/0 | 0/0 | 0/1 | 0/1 | 0/1 | 0/2 | 0/0 | 1/5 — Gender-specific event.
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 3
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3 | 0 | 0 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 4 | 2 | 1 | 2 | 11
Weight increased (Investigations) | 0 | 5 | 6 | 2 | 1 | 4 | 2 | 11
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 4 | 2 | 0 | 7 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 2 | 1 | 2 | 2 | 2 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 3
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Urethral discharge (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Penile blister (Reproductive system and breast disorders) | 0 | 0 | 0/19 | 0/19 | 0/19 | 0/18 | 1 | 0/58 — Gender-specific disorder
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/0 | 0/0 | 0/1 | 0/1 | 0/1 | 0/2 | 0/0 | 1/5 — Gender-specific disorder
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0/20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.